CLINICAL TRIAL: NCT07157748
Title: Effects of Compound Ejiao Syrup on Exercise Tolerance and Quality of Life in Critically Ill Patients After ICU Discharge: A Double-Blind, Multicenter,Randomized Controlled Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Tan Liang, Southwest hospital, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ThirdMMU-YCL
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Critically Ill Patients
Keywords: critically ill patients; exercise tolerance; exercise quality; Compound Ejiao Oral Liquid

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Fufang E'jiao Jiang (Experimental): Participants receive Fufang E'jiao Jiang, 20 mL orally three times daily for 90 days.
  Interventions: Drug: Fufang E'jiao Jiang
- Placebo Comparator: Matching Placebo (Placebo Comparator): Patients were given an equal-volume placebo (each vial containing compound Ejiao oral liquid [1 mL, 5%], caramel color [800 mg], and steviol glycosides [25 mg]) 20 mL orally, three times daily, for 90 consecutive days (identical to the compound Ejiao oral liquid in appearance, packaging, and taste).
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Fufang E'jiao Jiang — Oral solution; 20 mL TID for 90 days;
  Arms: Experimental: Fufang E'jiao Jiang
Drug: Matching Placebo — Oral solution; 20 mL TID for 90 days;
  Arms: Placebo Comparator: Matching Placebo

SUMMARY:
This study, titled "Effect of Compound Ejiao Jiang on Exercise Tolerance and Quality of Life of Critically Ill Patients after Discharge from ICU: A Double-Blind, Multicenter, Randomized Controlled Clinical Study (LIFT Study)," intends to enroll 156 patients (78 in the experimental group and 78 in the control group). A double-blind design will be adopted, with patients receiving Compound Ejiao Jiang (20 ml each time, three times a day for 90 consecutive days) or a placebo for intervention. The primary outcome measure is the 6-minute walking distance on the 90th day after randomization. Meanwhile, secondary endpoints such as physical function, quality of life, and nutritional and inflammatory indicators will also be monitored. The aim of this study is to explore the rehabilitation value of Compound Ejiao Jiang for patients with post-intensive care syndrome (PICS) through high-level evidence-based medicine methods and to provide scientific evidence for the integrated traditional Chinese and Western medicine approach to improving the long-term prognosis of critically ill patients

DETAILED DESCRIPTION:
This study aims to systematically evaluate the impact of the traditional Chinese medicine compound Ejiao Jiang on the long - term rehabilitation outcomes of critically ill patients after leaving the ICU through a rigorous double - blind, multi - center randomized controlled design, and provide scientific evidence for the improvement of the prognosis of critically ill patients through the combination of traditional Chinese and Western medicine. The following is a detailed breakdown of the protocol:

I. Basic Information of the Study Study Type: Multi - center, double - blind, randomized controlled trial. Study Period: From September 2025 to September 2027, covering the entire process of patient enrollment, follow - up, and data collation.

Sample Size: It is planned to include 156 eligible patients, who will be randomly assigned to the experimental group (78 cases) and the control group (78 cases) at a 1:1 ratio. The sample size calculation is based on the pre - experimental results of the primary endpoint (6 - minute walk distance).

II. Study Objectives

To evaluate the improvement effect of Ejiao Jiang on the exercise tolerance and quality of life of critically ill patients after leaving the ICU, specifically including:

Verify whether Ejiao Jiang can improve the patients' exercise tolerance (with the 6 - minute walk distance as the core indicator); Explore its impact on the patients' physical function, quality of life, nutritional status, and inflammatory response; Evaluate the safety of Ejiao Jiang during the critical illness rehabilitation period (such as the incidence of adverse reactions).

III. Screening of Study Subjects

1. Inclusion Criteria (Strictly Define the Target Population) Age: 18 - 75 years old (covering adult to elderly critically ill patients, excluding age - related extreme cases); Time Window: Within 24 hours after leaving the ICU (ensuring that the intervention starts in the early stage of rehabilitation, in line with the intervention timing of PICS); History of Critical Illness: Having received mechanical ventilation for ≥48 hours (indicating severe respiratory failure), and an ICU stay of 8 - 28 days (excluding patients with short - term mild illness or long - term dependence on the ICU); General Condition: Having started enteral nutrition (able to tolerate oral/tube feeding), spontaneous breathing (off mechanical ventilation), and clear consciousness (Glasgow Coma Scale, GCS ≥13 points); Exercise Ability: Being able to stand independently and complete the 6 - minute walk test (6MWT) (ensuring that the primary endpoint indicator can be measured).
2. Exclusion Criteria (Avoid Interfering Factors) Extremely Poor Prognosis: Expected to die within 48 hours or need to be readmitted to the ICU (unable to complete the follow - up); Severe Organ Dysfunction: Child - Pugh Class C (severe liver failure), creatinine clearance rate <40 mL/min (severe renal failure); Special Populations: Pregnant women and lactating women (to avoid the impact of the drug on the fetus/infant); Neurological/Psychiatric Diseases: Having a history of severe stroke, Parkinson's disease, schizophrenia, etc. (affecting the assessment of movement or cognition); Drug Conflict: Currently taking other traditional Chinese medicines for tonifying qi and nourishing blood (such as ginseng and astragalus preparations) (to avoid the superposition of traditional Chinese medicine components affecting the results).

IV. Design of Intervention Measures Experimental Group: Given Ejiao Jiang (specification: 20 ml/bottle), orally, 20 ml each time, 3 times a day, for 90 consecutive days (covering the critical period of critical illness rehabilitation, i.e., 3 months after leaving the ICU); Control Group: Given a placebo (with the same appearance and taste as Ejiao Jiang, prepared by a third - party institution), with the same usage and dosage as the experimental group;

Basic Treatment: Both groups of patients will receive a unified critical illness rehabilitation program, including:

Rehabilitation Guidance: 30 - minute bedside exercise, gait training, etc. every day; Nutritional Support: A personalized enteral nutrition plan will be developed according to the NRS - 2002 score; Regular Follow - up: A telephone follow - up once a week and an outpatient review once a month.

V. Outcome Indicator System (Comprehensively Evaluate the Rehabilitation Effect)

1. Primary Endpoint (Core Efficacy Indicator) 6 - Minute Walk Distance (6MWT): Measured on the 90th day after randomization to evaluate the patients' exercise tolerance.
2. Secondary Endpoints (Multi - dimensional Evaluation of Rehabilitation Outcomes) Physical Function: Including handgrip strength (muscle strength), gait speed (balance and coordination ability), Barthel Index (activities of daily living ability), and Fried Frailty Scale (frailty assessment); Quality of Life: The EQ - 5D - 5L questionnaire (European Quality of Life - 5 Dimensions - 5 Levels) will be used to evaluate the patients' self - perceived health (including 5 dimensions: mobility, self - care, usual activities, pain/discomfort, and anxiety/depression); Nutritional and Inflammatory Indicators: Laboratory tests of albumin (nutritional status), pre - albumin (short - term nutritional indicator), C - reactive protein (CRP, inflammatory response), procalcitonin (PCT, bacterial infection indicator), etc.; Clinical Outcomes: Mortality, readmission rate (to the ICU or general ward), non - hospitalized survival days (i.e., the number of days after discharge without readmission), etc.

ELIGIBILITY:
Inclusion Criteria:

* 1. Obtain informed consent; 2. Age between 18 and 75 years (inclusive); 3. Discharged from the ICU within 24 hours; 4. Received mechanical ventilation for at least 48 hours during this ICU stay; 5. Has been in the ICU for at least 8 days but no more than 28 days; 6. Enteral nutrition has been initiated. 7. Able to breathe spontaneously, with an oxygenation index (PaO2/FiO2) ≥ 200, and not requiring continuous high-flow oxygen therapy (e.g., nasal cannula flow ≤ 5 L/min); 8. Glasgow Coma Scale (GCS) score ≥ 13 at ICU discharge, and able to cooperate with study-related tests and follow-up; 9. Able to perform simple bedside activities with assistance (e.g., sitting up, standing, or short-distance walking); 10. No severe heart failure, no end-stage chronic respiratory failure, no lower-limb conditions that impair mobility, and no severe central nervous system disease; Able to stand independently and expected to complete the 6MWT at follow-up.

Exclusion Criteria:

* 1. Patients expected to die or for whom life-sustaining treatment will be withdrawn within 48 hours after ICU discharge; 2. Patients who need to be readmitted to the ICU within 1 week after ICU discharge; 3. Patients with persistent severe hepatic failure at ICU discharge (Child-Pugh class C); 4. Patients with persistent chronic kidney disease at ICU discharge (creatinine clearance < 40 mL/min); 5. Pregnant or breastfeeding patients; 6. Patients unable to walk independently before ICU admission (those who can walk independently with assistive devices may be included); 7. Traumatic brain injury, primary cerebrovascular diseases, brain tumors, or intracranial infections; 8. Primary cognitive impairment: Alzheimer's disease, vascular dementia, hydrocephalus, etc., and other serious central nervous system diseases; 9. History of psychiatric disorders such as depression, anxiety, or schizophrenia; 10. Occurrence of respiratory or cardiac arrest; 11. Patients with known cognitive impairment, lower-limb injury, systemic neuromuscular disease, or cranial/spinal conditions that could affect outcome assessment; 12. Patients currently taking other Qi- and blood-tonifying traditional Chinese medicines or patent Chinese medicines.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test (6MWT) | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital
  This evaluation is based on the walking distance that patients cover in six minutes when walking as fast as possible along a straight corridor, which is a indicator for assessing the lower limb motor function.

CONTACTS AND LOCATIONS:
Overall Officials: Changlin Yin, Ph,D, Principal Investigator — The First Affiliated Hospital of Army Medical University, Chongqing, China
Locations (1):
- the Southwest hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Ye T, Hong Z, Gong S, Zhou X, Liu H, Qian J, Qu H. Pharmacological and transcriptome profiling analyses of Fufang E'jiao Jiang during chemotherapy-induced myelosuppression in mice. J Ethnopharmacol. 2019 Jun 28;238:111869. doi: 10.1016/j.jep.2019.111869. Epub 2019 Apr 9. PMID 30978457
- [Background] Li Y, Zhang Z, Yang L, Li X, Zhou J, Li D, Luo S. Colla corii asini might upregulate ZNF471 and THOC5 by KRAB domain-containing zinc-finger protein pathway and THO complex subunit 5 pathway to improve anemia of pregnant women with beta-thalassemia. Ann Hematol. 2019 Aug;98(8):1813-1826. doi: 10.1007/s00277-019-03710-1. Epub 2019 May 16. PMID 31098739
- [Background] Li Y, He H, Yang L, Li X, Li D, Luo S. Therapeutic effect of Colla corii asini on improving anemia and hemoglobin compositions in pregnant women with thalassemia. Int J Hematol. 2016 Nov;104(5):559-565. doi: 10.1007/s12185-016-2069-0. Epub 2016 Jul 25. PMID 27456464
- [Background] Shi WB, Wang ZX, Liu HB, Jia YJ, Wang YP, Xu X, Zhang Y, Qi XD, Hu FD. Study on the mechanism of Fufang E'jiao Jiang on precancerous lesions of gastric cancer based on network pharmacology and metabolomics. J Ethnopharmacol. 2023 Mar 25;304:116030. doi: 10.1016/j.jep.2022.116030. Epub 2022 Dec 20. PMID 36563889
- [Background] Kress JP, Hall JB. ICU-acquired weakness and recovery from critical illness. N Engl J Med. 2014 Jul 17;371(3):287-8. doi: 10.1056/NEJMc1406274. No abstract available. PMID 25014703
- [Background] Iwashyna TJ, Ely EW, Smith DM, Langa KM. Long-term cognitive impairment and functional disability among survivors of severe sepsis. JAMA. 2010 Oct 27;304(16):1787-94. doi: 10.1001/jama.2010.1553. PMID 20978258
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Kaukonen KM, Bailey M, Suzuki S, Pilcher D, Bellomo R. Mortality related to severe sepsis and septic shock among critically ill patients in Australia and New Zealand, 2000-2012. JAMA. 2014 Apr 2;311(13):1308-16. doi: 10.1001/jama.2014.2637. PMID 24638143
- [Background] Pandharipande PP, Girard TD, Ely EW. Long-term cognitive impairment after critical illness. N Engl J Med. 2014 Jan 9;370(2):185-6. doi: 10.1056/NEJMc1313886. No abstract available. PMID 24401069
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660